CLINICAL TRIAL: NCT06007716
Title: The Effect Of Reflexology Massage On Pain, Anxiety And Comfort Level In Patients Undergoing Percutaneous Coronary Intervention
Brief Title: The Effect Of Reflexology On Pain, Anxiety And Comfort Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hakkari Universitesi (Other)
Responsible Party: Principal Investigator, Kamber Sumer, Assistant professor, Hakkari Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HU-SM-KM-01
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Myocardial Infarction; Angina Pectoris
MeSH Terms: conditions — Myocardial Infarction; Angina Pectoris | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: consists of experimental and placebo groups.
Who Masked: Participant
Masking Description: Participants were informed about the study after obtaining an informed consent form. It was noted that the participants had not received reflexology or classical massage before.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): it was planned to apply reflexology massage once a day for each patient for 2 consecutive days, in total 2 sessions.
  Interventions: Other: reflexology massage
- placebo group (Placebo Comparator): placebo massage was applied once a day for each patient for 2 consecutive days, for a total of 2 sessions.
  Interventions: Other: Placebo massage

INTERVENTIONS:
Other: reflexology massage — 5 minutes of classic message on the left foot, 15 minutes of reflexology message, and 5 minutes of classic message on the right foot, 15 minutes of reflexology message, a total of 40 minutes of massage. 30 minutes after the massage, evaluation was recorded with the Vital Signs Registration Form, McGill Pain Scale Short Form, State Anxiety Inventory, General Comfort Scale Short Form, and Fatigue and Quality Sleep Visual Comparison Scale. Thus, reflexology massage is performed once a day for each patient for 2 consecutive days, for a total of 2 sessions.
  Arms: Experimental group
Other: Placebo massage — Placebo reflexology massage was applied to each foot for 20 minutes, for a total of 40 minutes.30 minutes after the massage, evaluation was recorded with the Vital Signs Registration Form, McGill Pain Scale Short Form, State Anxiety Inventory, General Comfort Scale Short Form, and Fatigue and Quality Sleep Visual Comparison Scale. Thus, Placebo massage is performed once a day for each patient for 2 consecutive days, for a total of 2 sessions.
  Arms: placebo group

SUMMARY:
This study was performed as a randomized controlled a study with a pre test-post test design, aimed to determine affect of reflexology masagge to the pain, anxiety and comfort level on the patients that are percutaneous coronary intervention.

DETAILED DESCRIPTION:
A total of 74 patients, 37 in the experimental group and 37 in the placebo group, who met the criteria for inclusion in the study, constituted the sample of the study. Research data were collected with "Structured Patient Information Form", "Vital Signs Form", "State Anxiety Scale", "Visual Comparison Scale", "McGill Pain Scale Short Form" and "General Comfort Scale Short Form". Appropriate statistical methods were used in the analysis of the data.

Reflexology massage is a well tolerated, inexpensive, applicable and safe non-pharmacological method. The fact that nurses are educated and experienced about reflexology massage is of great importance for integrating reflexology massage into clinical settings.

If the results of this study are significant, it will be concluded that reflexology massage is effective in the management of pain and anxiety and increasing the comfort level in patients undergoing PCI. It will be recommended that reflexology massage be used in clinics to reduce pain, anxiety and increase comfort level in individuals undergoing PCI, and to include it in patient education. No study has been found in the national literature evaluating the effectiveness of reflexology massage in the management of PCI-related pain, anxiety and comfort. It is thought that this study will fill an important gap in the literature. The aim of this study, carried out in this context, is to reveal the effect of reflexology massage on pain, anxiety and comfort level in patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Literate, Diagnosed with PCI-related pain,
* Pain score of 4 out of 10 according to Visual Comparison Scale (VAS) after PCI.

Exclusion Criteria:

* Presence of a pacemaker,
* Having a diagnosis of diabetic foot,
* Presence of vision, hearing, cognitive ability impairment or psychosis,
* Being pregnant,
* Presence of disc herniation,
* Any contagious skin disease (shingles, fungus, etc.), open lesion/wound on the lower extremities, scar tissue, fracture, dislocation, amputation, edema, hematoma, thrombophlebitis, inflammatory and degenerative joint disease,
* Having applied reflexology massage in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The McGill Pain Scale Short Form-2 | 2 days
  The McGill Pain Scale Short Form, developed by Melzack in 1987, provides information about the sensory characteristics, severity and effect of pain. The validity and reliability study in Turkey was developed by Yakut et al. in 2007. McGill Pain Scale Short Form-2 (MAS-SF-2) was developed in 2010 by revising the McGill Pain Scale Short Form by Bicici and Günes.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | 2 days
  It was developed by Spielberger et al. in 1970 and validated and reliable in Turkish society by Öner and Le Compte (1977). The State-Trait Anxiety Inventory consists of two different parts and includes a total of 40 items, 20 of which are each.

OTHER OUTCOMES:
General Comfort Scale Short Form | 2 days
  General Comfort Scale Short Form GQS-SF was developed by Kolcaba in 2006. Validity and reliability were established by Saritas et al. in 2018. It includes the sub-dimensions of comfort, relief (9 items), relaxation (9 items), and overcoming problems (10 items).

CONTACTS AND LOCATIONS:
Overall Officials: Kamber SÜMER, Principal Investigator — PhD student
Locations (1):
- Van Regional Training and Research Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No